CLINICAL TRIAL: NCT04129970
Title: BITE: An Integrated Feasibility Trial and Case Series of Theta Burst Simulation in Binge Eating Disorder
Brief Title: Theta Burst Stimulation in Binge Eating Disorder: A Case Series
Acronym: BITE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID led to suspension of the study.New data suggest outcome measures should be revised and new approvals from research ethics committees will be needed
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pending Case Series
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2019-10

CONDITIONS: Binge-Eating Disorder
Keywords: Binge Eating; Transcranial Magnetic Stimulation; Theta Burst Stimulation; Neuromodulation; Psychiatric Disorders; Eating Disorders
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Mental Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Masking Description: All participants will receive active iTBS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent Theta Burst Stimulation (Experimental): The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer active iTBS.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — iTBS will be delivered to the left dorsolateral prefrontal cortex (DLPFC) at 80% of resting motor threshold using standard stimulation parameters; triplet-bursts will be delivered at high frequency (50 Hz) with an inter-burst interval of 200 ms. Each TBS train will last 2 seconds and consists of 10 triplet-bursts (30 pulses). Each iTBS session will involve 10 TBS trains repeated every 10 seconds for 190 seconds, with a total number of 600 pulses delivered during each session.
  Other Names: iTBS

SUMMARY:
Binge eating disorder (BED) is a common and disabling eating disorder (ED) which presents a substantial disease burden. Individuals seeking treatment for binge eating difficulties typically receive talking therapy treatment however, treatment response is inadequate. As such, it is imperative that novel treatment options be identified.

Repetitive transcranial magnetic stimulation (rTMS) techniques are well established for the treatment of depression and preliminary findings indicate that similarly therapeutic effects may occur in populations with eating difficulties. Intermittent theta burst stimulation (iTBS) is a novel variant of excitatory rTMS which is emerging as an attractive alternative to standard stimulation. This trial aims to assess the feasibility of conducting a large scale randomised controlled trial (RCT) investigating theta burst in individuals with binge eating disorder, and to examine whether theta burst stimulation may improve symptoms in this population.

DETAILED DESCRIPTION:
Binge eating is a common and disabling problem which is often associated with obesity. Binge eating causes significant distress and compromises quality of life in affected individuals. Current treatments do not support full recovery in a considerable number of adults and adolescents. As such, it is important that we explore new options for treatment.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive procedure that is emerging as a potentially effective treatment psychiatric disorders. In rTMS, an electric current is passed through a coil placed on the scalp. This current creates a magnetic field which changes the activity in the brain area immediately below. rTMS is a well-established treatment for depression and has been approved by the National Institute for Care and Excellence (NICE; 2015). The NICE-approved rTMS treatment for depression involves 20-30 sessions, each requiring 37.5 minutes of stimulation. A novel variant of rTMS, intermittent theta burst stimulation (iTBS), is an attractive alternative to standard stimulation which is delivered using a very similar procedure as standard rTMS and may produce comparable effects in as little as 3 minutes.

In depression, the therapeutic applications for rTMS have been widely studied. By comparison, research in eating disorders and obesity are preliminary. Nevertheless, studies have reported promising results in these populations. For example, a case study involving a patient with refractory BED and comorbid depression reported clinical improvement following 20 sessions of high frequency (excitatory) rTMS targeting the left DLPFC (Baczynski et al, 2014). Similarly, two recent studies of obese adults have reported a reduction in food intake, reduced craving, and significant weight loss following 20 sessions of high frequency rTMS targeting the left DLPFC (Alvarado-Reynoso & Ambriz-Tututi, 2019; Kim et al, 2018). Finally, studies in healthy participants reporting strong cravings and clinical participants with bulimia nervosa have also reported a reduction in craving and food-intake following high frequency rTMS (for example, Dunlop et al, 2015; Van den Eynde, 2010, and Uher et al, 2010). No study to date has used iTBS in eating disorders.

The primary objective for this trial is to assess whether iTBS may benefit people with binge eating difficulties. As such, we are conducting two inter-related studies: (1) a proof-of-concept randomised double-blind sham-controlled trial involving a single-session of either real or sham iTBS, and (2) a therapeutic case series involving 20 sessions of real iTBS delivered week-daily over four consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* Meets DSM-5 criteria for full-syndrome BED
* Overweight or obese according to World Health Organisation (WHO) criteria (BMI>25 kg/m2 for adults, and a weight-for-height greater than 2 standard deviations above the median for adolescents).

Exclusion Criteria:

* All known contraindications to MRI and TBS (assessed using TMS and MRI safety screening questionnaires)
* Pregnancy (or suspected pregnancy)
* History of neurological disease and/or seizure
* Having any metallic implants anywhere in the head or body
* History of head or eye injury; significant health problems in the previous six months;
* Lifetime diagnosis of substance dependence, psychosis, bipolar disorder, borderline personality disorder
* Other primary psychiatric disorder requiring treatment in its own right
* Taking psychotropic medication other than a stable dosage of selective serotonin reuptake inhibitors (SSRI) for at least 14 days prior to study enrollment
* Alcohol consumption exceeding 14 units per week
* Cigarette consumption or nicotine replacement exceeding >15 cigarettes daily or equivalent.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Core symptoms of BED | Baseline to 3 months post-iTBS
  An index of BED symptoms will be computed by summing the scores on four 10cm visual analogue scales (VAS) assessing levels of current hunger, craving for food, urge to eat and urge to binge eat. Change in BED symptoms will be assessed to determine whether iTBS may affect core symptoms of BED.
Global EDE-Q Score | Baseline to 3 months post-iTBS
  The EDE-Q is a 28-item questionnaire that provides a measure of the range and severity of eating disorder features experienced over the past 28 days. Change in the EDE-Q Global score will be used to determine whether iTBS may affect BED diagnosis and/or severity.

SECONDARY OUTCOMES:
Negative Affect as measured by the DASS-21 | Baseline to 3 months post-iTBS
  The DASS-21 will be used to determine whether iTBS may alter negative affect in participants with BED. The DASS-21 is a self-report questionnaire of 21 items, 7 items per sub-scale: depression, anxiety and stress.
Trait Level Craving for Food | Baseline to 3 months post-iTBS
  The Food Craving Questionnaire (FCQ, Trait) is a 15 item, self-report questionnaire that measures trait levels of craving for food across 9 domains. The FCQ will be used to examine whether iTBS may effect trait-level craving for food in participants with BED.
Eating Disorder Related Clinical Impairment | Baseline to 3 months post-iTBS
  The Clinical Impairment Assessment (CIA) is designed to assess quality of life by exploring the perceived effects of having an ED on various domains, including social, emotional and cognitive aspects. The CIA will be used to assess whether participants report a change in their ED related quality of life following 20-sessions of iTBS.
Body Mass Index | Baseline to 3 months post-iTBS
  Weight in kilograms(kg) and height in metres(m) will be combined to report BMI in kg/m^2 to determine whether 20 sessions of iTBS may be associated with change in BMI.
Body Fat | Baseline to 3 months post-iTBS
  Body fat, derived by Bioelectrical Impedance Analysiso, will be used to determine whether iTBS is associated with a change in body composition.
Delay Discounting | Baseline to 3 months post-iTBS
  To determine whether iTBS may improve study self-regulation, delayed gratification and valuation of reward, change in performance on the delay discounting task will be assessed.
Emotion Regulation | Baseline to 3 months post-iTBS
  To determine whether iTBS may alter emotion regulation we will assess whether, following 20-sessions of iTBS, there is a change in heart rate variability while viewing the International Affective Picture System.
Food Choice | Baseline to 3 months post-iTBS
  To determine whether iTBS may alter food-related decision making participants will perform a neuropsychological task measuring decision making regarding food selection prior to and following iTBS treatment, and at 3 month follow up.
Inhibitory Control | Baseline to 3 months post-iTBS
  The cued go/no go task is a useful measure of impulse control in clinical populations. This task is a classic test of executive function, requiring effortful response inhibition. To determine whether iTBS may alter impulse control participants will perform a cued go/no go task prior to and following iTBS treatment, and at 3 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Schmidt, Principal Investigator — King's College London
Locations (1):
- King's College London Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No